CLINICAL TRIAL: NCT01225523
Title: Perioperative Versus Preoperative Chemotherapy With Surgery in Patients With Locoregional Squamous Carcinoma of Esophagus
Brief Title: Perioperative Vs. Preoperative Chemotherapy With Surgery in the Squamous Carcinoma of Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZY-01
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-09

CONDITIONS: Squamous Carcinoma of Esophagus; Esophagus Disorders
MeSH Terms: conditions — Esophageal Diseases | interventions — Paclitaxel; Cisplatin; Fluorouracil; Capecitabine

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Preoperative chemotherapy followed by surgery (Active Comparator)
  Interventions: Drug: Paclitaxel; Cisplatin; 5-Fluorouracil
- Perioperative chemotherapy with surgery (Active Comparator)
  Interventions: Drug: Paclitaxel; Cisplatin; 5-Fluorouracil; Drug: Paclitaxel; Cisplatin; 5-Fluorouracil; Capecitabine

INTERVENTIONS:
Drug: Paclitaxel; Cisplatin; 5-Fluorouracil — Two preoperative cycles with Paclitaxel 200 mg/m² d1, Cisplatin 60 mg/m² d1, 5-Fluorouracil 700 mg/m² d1-5 repeated every 3 weeks followed by resection
Drug: Paclitaxel; Cisplatin; 5-Fluorouracil; Capecitabine — Two postoperative cycles with Paclitaxel 200 mg/m²/day d1, Cisplatin 60 mg/m²/day d1, 5-Fluorouracil 700 mg/m²/day d1-5 repeated every 3 weeks Among patients with no responses to preoperative chemotherapy, Capecitabine 625 mg/m² twice-daily dose as alternatives to infused 5-Fluorouracil in the postoperative chemotherapy regimen
  Arms: Perioperative chemotherapy with surgery

SUMMARY:
To assess whether or not a perioperative therapy with surgery can improve the outcomes among patients with potentially curable squamous carcinoma of esophagus as compared to a preoperative chemotherapy followed by surgery

DETAILED DESCRIPTION:
Perioperative chemotherapy has been shown to significantly improve the R0 resection rate, the disease free survival and the overall survival in patients with adenocarcinoma of the esophagus, the gastroesophageal junction and the stomach. Therefore, perioperative chemotherapy is the new therapeutic standard (Cunningham NEJM 2006, MRC, Lancet 2002, Boige ASCO 2007). The best-evaluated regime is the combination of Epirubicin, Cisplatin and 5-FU (ECF) (Cunningham, NEJM 2007). Cisplatin and 5-FU are considered to be the most important components to form the cornerstone of this regime.

Paclitaxel is a new and highly active cytotoxic agent. In a randomized phase II study, the dual combination of Paclitaxel and 5-FU seemed to show similar effects as ECF, administered as first line treatment. The triplet combination of Paclitaxel, Cisplatin and 5-FU has significantly superior efficacy than a combination of Cisplatin und 5-FU (Van Cutsem, JCO 2007).

It has been shown that Capecitabine is more active than 5-FU and can replace intravenous 5-FU in the combination with Cisplatin in the treatment of esophageal cancer. Capecitabine therefore is FDA approved for esophageal cancer (Cunningham, ASCO 2006, Kang ASCO 2006).It seems reasonable to optimize perioperative chemotherapy by including this modern chemotherapeutics.

In this study, patients with squamous carcinoma of esophagus and gastroesophageal junction who seem operable with curative intent according to oncological and surgical assessment are treated with 2 preoperative cycles of PCF followed by surgical resection, followed by 2 postoperative cycles of PCF. Among patients with no responses to preoperative chemotherapy, Capecitabine 625 mg/m² twice-daily dose is defined as alternatives to infused 5-Fluorouracil in the postoperative chemotherapy regimen Postoperative chemotherapy will start within 4-6 weeks after the operation. 3 weeks after the end of the last chemotherapy the final investigation (end of study visit) will be done.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* histologically confirmed esophageal cancer (squamous carcinoma) measurable, non-metastatic disease
* no previous cancer therapy (chemotherapy, radiotherapy or resection)
* life expectancy > 3 months
* age > 18 years
* WHO Status ≤ 1
* Intended curative resection according to evaluation of an experienced surgeon
* Negative pregnancy blood test at screening but not earlier than 72 hours prior to start of chemotherapy for women with child bearing potential
* Adequate haematologic function and liver and renal function: neutrophils > 1.5×109/L; thrombocytes > 100×109/L; haemoglobin > 10 g/dl, creatinine clearance > 60 ml/min (calculated according to Cockroft and Gault), total bilirubin < 1.0×UNL; AST and ALT < 1.5×UNL, AP < 2.5×UNL
* Complete staging within 3 weeks prior to start of treatment (CT-scan of thorax and abdomen, endosonography, gastroscopy)
* Ability to keep appointments and follow the study protocol
* By CT-scan, endoscopy or endosonography measurable or evaluable disease

Exclusion Criteria:

* Former therapy of cancer (operation, chemo- or radiotherapy)
* Diagnosis of another cancer in the last 5 years prior to study entry which has not been cured by operation only (exception in-situ-carcinoma of the cervix or cured non-melanomatose skin cancer)
* Known contraindication to the planned chemotherapeutics
* Presence of distant metastases
* Anamnestic known serious disease or other concomitant diseases that affect participation in this study, such as:

oInstable cardiac disease: symptomatic heart failure, symptomatic coronary artery disease, ventricular cardiac arrhythmia not well controlled with medication, myocardial infarction or resuscitation within 6 month before study oActive infection necessitating systemic therapy or uncontrolled infection oInterstitial lung diseases (for example: pneumonitis or fibrosis of the lung) and indication for interstitial lung disease in chest x-ray or CT-scan respectively oActive inflammatory bowel disease or other bowel diseases which provoke chronic diarrhea (defined as > 4 bowel movements per day) oNeurological or psychiatric disease including dementia, epilepsy or untreated, symptomatic brain metastases oLimited hearing ability

* Presence of upper GI obstruction, leading to inability to swallow ground tablets
* Presence of acute or chronic systemic infection
* Presence of a bowel obstruction within the last 30 days
* Pregnant or lactating women or women with child bearing potential and men without adequate contraception (high effective contraception, defined as Pearl Index < 1) like birth control pill, hormone spiral, hormone implant, transdermal patch, a combination of two barrier methods (condom and diaphragm), realized sterilization or sexual abstinence during the study and at least for 3 months after the last infusion
* Any other situation which may lead to an unacceptable high risk for the patient, when he participates in the study
* Parallel treatment in another clinical study or prior participation in this study
* Treatment with any other therapy against the tumor or any parallel radiation
* Symptomatic peripheral neuropathy NCI-CTCAE degree > 2
* Intolerance to the study medication
* Detention in a psychiatric unit or imprisonment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 1997-01; Primary Completion 2008-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 5 years
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Pathological remission rate | After 2 cycles of preoperative chemotherapy (2 month)
Resectability rate | After 2 cycles of preoperative chemotherapy (2 month)
Operative and postoperative complication rate | Within 30 days after surgery
30-day mortality | After date of surgery
Toxicity of preoperative and postoperative chemotherapy
Rate of local recurrences and metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of College of Medicine of Xi'an Jiao Tong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zhao Y, Dai Z, Min W, Sui X, Kang H, Zhang Y, Ren H, Wang XJ. Perioperative versus Preoperative Chemotherapy with Surgery in Patients with Resectable Squamous Cell Carcinoma of Esophagus: A Phase III Randomized Trial. J Thorac Oncol. 2015 Sep;10(9):1349-1356. doi: 10.1097/JTO.0000000000000612. PMID 26287319